CLINICAL TRIAL: NCT05944913
Title: Randomized Study Comparing Negative Pressure Dressing Versus Conventional Dressing in Patients With Resected Limb or Trunk Soft Tissue Sarcoma (STS) After External Radiotherapy
Brief Title: Study Comparing Negative Pressure Dressing vs Conventional in Patients With Resected STS After Radiotherapy
Acronym: TPN-RAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ET22-146
Record Dates: First submitted 2023-06-26; First posted 2023-07-13 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Soft Tissue Sarcoma
Keywords: STS; Negative Pressure Wound Therapy; Surgery with preoperative irradiation
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Intervention Model Description: The randomization (1:1 ratio) will be stratified according to STS location (upper limb vs lower limb vs trunk) and ASA class (1 or 2 vs ≥ 3).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A : Surgery for STS and prevena (Experimental): The surgery for the STS lesion will be performed according to standard practices.
  PREVENA™ Incision Management System should be applied immediately post-surgery to clean surgically closed wounds. It should be continuously applied for a minimum of 2 days and up to a maximum of 7 days (as per PREVENA user manual)
  Interventions: Device: Prevena
- Arm B : Surgery for STS and standard postoperative wound management (No Intervention): The surgery for the STS lesion will be performed according to standard practices.
  The dressing and drainage of the wound will be performed according to usual practices, with the exception of negative pressure dressings.

INTERVENTIONS:
Device: Prevena — PREVENA™ is a CE-marked class IIa medical device. The PREVENA™ Incision Management System is also intended to manage the environment of closed surgical incisions and surround intact skin in patients at risk for developing post-operative complications, such as infection, by maintaining a closed environment via the application of a negative pressure wound therapy system to the incision.
  Arms: Arm A : Surgery for STS and prevena

SUMMARY:
This is a randomized (1:1 ratio), prospective, comparative, controlled, open-label study. The aim is to compare the efficacy of negative pressure therapy (PREVENA™) versus standard postoperative wound management on the wound healing after surgery for previously irradiated Soft Tissue Sarcoma (STS)

DETAILED DESCRIPTION:
The gold standard treatment for primary non-metastatic STS is complete surgical resection. Peri-operative Radiation Therapy (RT) has been proved to improve local control . Nevertheless, the timing of RT, whether preoperative or postoperative, remains a debate.

Both have similar local control efficacy, but preoperative RT results in lower rates of long-term fibrosis and lymphedema and improved joint mobility than postoperative RT. On the other hand, the adverse effect of pre-operative RT is a higher rate of wound post-operative complications and re-operations.

Any effort to reduce the high rate of postoperative complications could offer the advantage of preoperative RT in terms of reduced long-term sequelae compared with postoperative RT without a higher wound complication rate postoperatively. Short retrospective series of Negative Pressure Wound Therapy (NPWT) after surgical resection of Soft Tissue Sarcoma (STS) have reported very encouraging results in preventing wound complications: patients treated with NPWT were less likely to develop wound complications than those who did not receive it. Both groups did not report an increased rate of local recurrence. The use of NPWT would also reduce the cost of care by avoiding complications.

That's why the investigators propose this study comparing the use of a negative pressure dressing to a conventional dressing in patients with STS of the limbs or trunk resected after neo-adjuvant external radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the day of consenting to the study
* Patients with primary STS of the limb or trunk treated with preoperative external radiation therapy (decided in multidisciplinary board)
* Intent to cure resection required for STS planned between 3 to 8 weeks after the end of RT
* Planned primary wound closure, including local or distant jambeau
* Ability to understand and willingness for follow-up visits
* Covered by a medical insurance
* Signed and dated informed consent document indicating that the patient has been informed of all aspects of the trial prior to enrolment.

Exclusion Criteria:

* Known hypersensibility to silver
* Patients with a diagnosis of Ewing's sarcoma, chondrosarcoma, osteosarcoma, or desmoid tumor. Nota bene: Only patients with bone tumors are affected; patients with soft tissue tumors can be included in the study.
* Patient in relapse setting;
* Patient requiring a surgical revision after R1 or R2 resection;
* Planned blade drainage;
* Planned no wound-closure and skin graft after resection
* Patient requiring authorship or curators or patient deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2023-08-03 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
The efficacy of negative pressure therapy (PREVENA) versus standard postoperative wound management on the wound healing after surgery for previously irradiated STS | Within the 3-month postoperative period.
  Assessed by major wound complications rate

SECONDARY OUTCOMES:
Three month deep infection rate | At 3 months post-surgery visit
  Assessed by the proportion of patients experiencing a second surgery for wound healing problem within 3 postoperative months
Three months secondary surgery for wound healing problem rate | At 3 months post-surgery visit
  Assessed by the proportion of patients experiencing a second surgery for wound healing problem within 3 postoperative months
Hospitalization duration | At 3 months post-surgery visit
  Defined as the number of hospitalization days from the date of surgery to the date of discharge
Time to complete wound healing | Up to 27 months
  Defined as the interval from surgery to 100% healing (total wound closure with no need for dressing and any local care)
Number and types of major wound complications (MWCs) | Up to 27 months
  Assessed by a number and differens types of a major wound complications
Quality of life using EQ-5D-5L | At 28 days and 3 months after surgery for each patients
  Assessed by EQ-5D-5L introduce by EuroQol Group in 2009 with five dimensions : mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has five levels : no problems, slight problems, moderate problems, severe problems and extreme problems. A minimum value is 0 and a maximum value is 100. A mean worst value is 0 and a better mean value is 100.
Incidence of Adverse Events | Up to 27months
  Defined by the number of patients with Adverse Events (any type and any grade using the NCI-CTC AE scale version 5.0)
Quality of life using FACT-G | At 28 days and 3 months after surgery for each patients
  Assessed by FACT-G : Functionnal Assesment of Cancer Therapy with 27 items. There are four domains of HRQOL in cancer patients: Physical, social, emotional, and functional well-being. A minimum value is 0 and a maximum value is 4. A mean worst value is 0 and a better mean value is 108.

CONTACTS AND LOCATIONS:
Overall Officials: François Gouin, MD, Chirurgien, Principal Investigator — Centre Leon Berard
Locations (15):
- France (15):
  - CHU Nantes, Nantes, Pays de Loire
  - Centre Leon Berard, Lyon, Rhône-Alpes Auvergne
  - Institut de Cancérologie de l'Ouest - Pays de Loire, Angers
  - Institut Bergonié, Bordeaux
  - CHRU Tours Hôpital Trousseau, Chambray-lès-Tours
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar Lambert, Lille
  - CHU Limoges, Limoges
  - Institut du Cancer de Montpellier, Montpellier
  - Institut Curie, Paris
  - APHP Hôpital Cochin, Paris
  - CHU Rennes, Rennes
  - IUCT Oncopole, Toulouse
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy